CLINICAL TRIAL: NCT02705456
Title: Enamel Caries in Orthodontic Patients
Acronym: ECOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: University Hospital Regensburg (Other); University Hospital Munich (Other); University Hospital Dresden (Other); Goethe University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ulrich Schlagenhauf, Chairman Dept. of Periodontology, Wuerzburg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ECOP1
Record Dates: First submitted 2016-02-25; First posted 2016-03-10 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Dental Caries
Keywords: Dental Caries; Tooth Paste; Orthodontics; Fluorides
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HA-Tooth Paste (Experimental): Tooth Brushing HA
  Cleaning of all teeth using a standardized electric tooth brush and a non-fluoridated tooth paste containing microcrystalline hydroxylapatite twice daily over the duration of the study (24 weeks).
  Professional caries prevention by professional supragingival tooth cleaning and the subsequent application of a 1% chlorhexidine gel once every 4 weeks over the duration of the study (24 weeks).
  Interventions: Procedure: Tooth Brushing HA
- FL-Tooth Paste (Active Comparator): Tooth Brushing FL
  Cleaning of all teeth using a standardized electric tooth brush and a fluoridated tooth paste twice daily over the duration of the study (24 weeks).
  Professional caries prevention by professional supragingival tooth cleaning and the subsequent application of a 1% chlorhexidine gel once every 4 weeks over the duration of the study (24 weeks).
  Interventions: Procedure: Tooth Brushing FL

INTERVENTIONS:
Procedure: Tooth Brushing HA — 2x daily repeated cleaning of all teeth using a standardized electric tooth brush and a non-fluoridated tooth paste containing microcrystalline hydroxylapatite.
  Professional supragingival tooth cleaning once every 4 weeks with a rubber cup followed by the application of a 1% chlorhexidine gel over the duration of the study (24 weeks).
  Arms: HA-Tooth Paste
Procedure: Tooth Brushing FL — 2x daily repeated cleaning of all teeth using a standardized electric tooth brush and a fluoridated tooth paste.
  Professional supragingival tooth cleaning once every 4 weeks with a rubber cup followed by the application of a 1% chlorhexidine gel over the duration of the study (24 weeks).
  Arms: FL-Tooth Paste

SUMMARY:
This randomized double-blind two arm controlled clinical trials evaluates the hypothesis that the regular use of a tooth paste containing microcrystalline hydroxylapatite provides a caries preventive effect in caries-susceptible individuals undergoing orthodontic therapy with fixed appliances which is comparable to the caries preventive effect provided by the regular use of a fluoridated tooth paste.

DETAILED DESCRIPTION:
Introduction

According to the criteria of evidence based medicine the use of fluoridated tooth paste as well as fluoridated mouth rinses are,with the exception of dietary control, the only proven measures for the prevention of dental caries.

Aim, Study Hypothesis

The aim of this randomized double-blind, two arm, controlled clinical trial is evaluation of the hypothesis that the regular use of a tooth paste containing microcrystalline particles of hydroxylapatite in caries-active subjects under orthodontic therapy with fixed appliances will provide at least a comparable extent of caries prevention as the regular use of fluoridated tooth paste during an observation period of 6 months.

Material and Methods

Study subjects will be recruited from juveniles and young adults, age 12-25, displaying high (≥105 CFU) salivary counts of caries promoting mutans streptococci and seeking orthodontic therapy with fixed appliances. Evaluated parameters are the presence of enamel caries on the buccal aspects of teeth 15-25 according to the criteria of the International Caries Detection and Assessment System (ICDAS), the presence of gingival inflammation assessed by the Gingival Index (GI) the presence of microbial plaque on the evaluated teeth assessed by the Plaque Index (PlI) and the extent of mutans streptococci colonization (MS) on the evaluated teeth and in saliva using standardized cultivation techniques. Primary endpoint of the study is the number and severity of enamel caries lesions according to the ICDAS classification. Exclusion criteria are the presence of ICDAS lesion ≥ 3 on the buccal surfaces of teeth 15-25, the presence of gingival lesions > GI 2 and the regular use of salivary flow-reducing medications.

At baseline, ICDAS scores, as well as GI, PlI and MS will be recorded followed by the incorporation of the fixed orthodontic appliances. Subsequently, using a random list participants are provided with a standardized electric tooth brush and a supply of one of the two experimental tooth pastes (hydroxylapatite(HA)/fluoride (FL)) to be used 2 x daily for the next 6 months. HA-tooth paste contains no fluoride, FL-tooth paste contains stannous fluoride and amine fluoride. At days 28, 84 and 168 (end of study) ICDAS, GI, PlI and MS are recorded again. Additionally all study participants will receive a full mouth preventive professional supragingival tooth cleaning followed by the application of a 1% chlorhexidine gel on all tooth surfaces once every 4 weeks during the course of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy juveniles and young adults with caries-promoting mutans streptococci colonization seeking orthodontic therapy with fixed orthodontic appliances

Exclusion Criteria:

* Oral ulcers
* Caries lesions on the buccal aspects of teeth 15-25
* Unrestored caries on any tooth
* Regular use of medications interfering with salivary flow and/or gingival inflammation

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2014-10; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of developing enamel caries lesions | 168 days (24 weeks)
  Recording of newly developing enamel caries lesions according to the International Caries Detection and Assessment System (ICDAS)

SECONDARY OUTCOMES:
Gingival Inflammation using the Gingival Index | 168 days (24 weeks)
  Assessment of gingival inflammation using the Gingival Index
Plaque Coverage using the Plaque Index | 168 days (24 weeks)
  Assessment of bacterial plaque coverage using the Plaque Index (Silness u. Loe 1964)
Mutans Streptococci Colonization | 168 days (24 weeks)
  Assessment of mutans streptococci colonization in saliva and on tooth surfaces

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schlagenhauf, Prof. Dr., Principal Investigator — Wuerzburg University Hospital
Locations (1):
- Dept. of Periodontology, University Hospital Wuerzburg, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schlagenhauf U, Kunzelmann KH, Hannig C, May TW, Hosl H, Gratza M, Viergutz G, Nazet M, Schamberger S, Proff P. Impact of a non-fluoridated microcrystalline hydroxyapatite dentifrice on enamel caries progression in highly caries-susceptible orthodontic patients: A randomized, controlled 6-month trial. J Investig Clin Dent. 2019 May;10(2):e12399. doi: 10.1111/jicd.12399. Epub 2019 Jan 30. PMID 30701704